CLINICAL TRIAL: NCT06743308
Title: Information Needs, Preferences, and Understanding Trial (INPUT): A Randomized, Controlled Trial of the Effects of a Screening Tool on Illness Understanding
Brief Title: Novel INPUT Screening Tool to Improve Illness Understanding in Patients With Metastatic or Incurable Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1519; NCI-2024-10305 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Lung Carcinoma; Metastatic Lung Carcinoma; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Masking Description: The research staff conducting the outcomes assessment (other than acceptability) will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Standard care) (Active Comparator): Patients undergo standard of care oncology follow-up visits.
  Interventions: Other: Best Practice; Other: Questionnaire Administration
- Arm II (INPUT screening) (Experimental): Patients complete the INPUT screening tool at each of their standard of care follow up visits, with their medical oncology team.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Other Best Practice best practice, standard of care, standard of care, standard of care, standard therapy Undergo standard of care oncology follow-up visits
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial compares the use of a new screening tool designed to evaluate patients' information needs, preferences, and illness understanding to the usual care to improve illness understanding in patients with lung cancer that has spread from where it first started (primary site) to other places in the body (metastatic) or for which no curative treatment is currently available (incurable). Goal concordant care is a model of care that aligns a patient's medical care with their values, preferences, and goals. Often, patients may not fully understand their illness and prognosis, but this information is important so that they can make fully informed decisions regarding their care that are consistent with their values, preferences, and goals. Completing the Information Needs, Preferences, and Understanding Trial (INPUT) screening tool may allow for more frequent and regular discussions regarding disease status and treatment goals, ultimately resulting in improved patient illness understanding and goal concordant care for patients with metastatic or incurable lung cancer.

DETAILED DESCRIPTION:
Primary Objectives To estimate the within group effect of perception of curability over 3 months in both the systematic screening group and the usual care group among patients with metastatic or incurable lung cancer who present to the thoracic medical oncology clinic at The University of Texas MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Within 3 months of biopsy-confirmed diagnosis of stage IV lung cancer
* Age 18 or over
* English speaking
* Attending a follow-up visit at the thoracic medical oncology clinic
* Plans to receive or actively undergoing cancer-directed systemic treatment at MD Anderson

Exclusion Criteria:

• Diagnosis of cognitive impairment or dementia requiring a surrogate decision maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in illness understanding | At 3 months
  Binary curability status is derived from the response to the INPUT Screening survey question #2. Will be similarly modeled by mixed-effect logistic regression.

SECONDARY OUTCOMES:
Difference between treatment groups in illness understanding | At 3 and 6 months
  Based upon the Prigerson Measure of Illness Understanding. The Likert-scale and composite score responses (excluding the acceptability of screening tool assessment) will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts.
Quality of communication | At 3 and 6 months
  Assessed via the Quality of Communication questionnaire. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Feeling heard and understood by healthcare team | At 3 and 6 months
  Assessed via the Feeling Heard and Understood scale. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Death-related anxiety | At 3 and 6 months
  Assessed via the Death and Dying Distress scale. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Anxiety related symptoms | At 3 and 6 months
  Assessed via the Generalized Anxiety Disorder scale. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Depression | At 3 and 6 months
  Assessed via the Patient Health Questionnaire, 9 items. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Health related quality of life | At 3 and 6 months
  Assessed via the Functional Assessment of Cancer Therapy - General. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Symptoms of advanced cancer | At 3 and 6 months
  Assessed via the Edmonton Symptom Assessment System. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.
Acceptability of screening tool | At 3 months
  Assessed via the Ease of Use, Acceptability, Usefulness, and Safety questionnaire.
Goals of care | At 3 and 6 months
  Assessed via Goals of Care. The Likert-scale and composite score responses will be modeled by mixed-effect analysis of variance with relation to treatment group and time point, with interaction. Change from baseline at each time point will be assessed by contrasts, without adjustment for multiple comparisons since this is a pilot study. Baseline variables which show evidence of differences may be utilized as model covariates to control for associated bias. Binary responses (including the primary objective) will be similarly modeled by mixed-effect logistic regression. Survey responses which are neither Likert, composite, nor binary, may have categories collapsed such that they can be analyzed as binary.

CONTACTS AND LOCATIONS:
Overall Officials: Kayley Ancy, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org